CLINICAL TRIAL: NCT06401382
Title: The Impact of A Modified Aligner Appliance With NiTi Springs and Conventional Fixed Appliances on Oral Health-related Quality of Life in Patients With Mild Crowding
Brief Title: Oral Health-Related Quality of Life Between Two Different Types of Orthodontic Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-2-2024
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified aligner appliance with NiTi springs (Experimental): The patients in this group will be treated using a Modified aligner appliance with NiTi springs.
  Interventions: Device: A modified aligner appliance with NiTi springs
- Conventional fixed appliances (Active Comparator): The patients in this group will be treated using conventional fixed appliances.
  Interventions: Device: Conventional fixed appliances

INTERVENTIONS:
Device: A modified aligner appliance with NiTi springs — The modified aligner appliance will be used until the final position is achieved.
  Arms: Modified aligner appliance with NiTi springs
Device: Conventional fixed appliances — The traditional fixed appliances with a standard prescription will be used.
  Arms: Conventional fixed appliances

SUMMARY:
Patients who have mild crowding from the Orthodontic Department at University of Damascus Dental School will be treated in this trial. The effects of modified aligner appliance with NiTi springs on oral health-related quality of life (OHRQoL) compared with conventional fixed appliances using the OHIP-14 questionnaire during orthodontic treatment. So, this study aims to compare the changes in OHRQoL between patients receiving modified aligner appliances or conventional fixed appliances during orthodontic treatment.

There are two groups:

1. Experimental group: the patients in this group will be treated using a modified aligner appliance.
2. Control group: the patients in this group will be treated using conventional fixed appliances

DETAILED DESCRIPTION:
Most adult patients do not choose traditional fixed appliances due to concerns about appearance, lengthy treatment time, and challenges with oral hygiene. This study aimed to assess the impact on psychological well-being, aesthetics, and functionality of a novel single aligner appliance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between (18 - 25) years.
2. Mild crowding < 4 mm in the lower dental arch with class I malocclusion
3. No congenitally missing or extracted teeth (except for third molars)
4. Patients with good oral hygiene.

Exclusion Criteria:

1. Bimaxillary dentoalveolar protrusion.
2. Previous orthodontic treatment.
3. Severe skeletal discrepancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Changes in oral health related quality of life | T0: immediately before the start of orthodontic treatment; T1: after two weeks; T2: after one months; T3: after two months; T4: post-treatment
  Patients in both groups will receive a survey called the Oral-Health-Impact-Profile with 14 items (OHIP-14) to complete at every adjustment visit. The OHIP-14 questionnaire assesses various aspects of the individual's oral health, functional well-being, emotional well-being, expectations, and satisfaction with care, and sense of self through subjective evaluation. The total score can range from 0 to 56, with higher scores indicating poorer OHRQoL. Each domain within the OHIP-14 score is also rated on a scale of 0 to 8, with individual items contributing a score of 0 to 4.

SECONDARY OUTCOMES:
Patient satisfaction with the progress of the treatment | At the end of treatment which is expected to occur within 4 to 6 months
  Patients in both groups will be asked one question about their satisfaction with the treatment's progress. This question records satisfaction using a 100 mm visual analog scale (VAS). The left end of the line refers to no satisfaction (VAS=0), whereas the right end refers to maximum satisfaction (VAS=100).
Patient satisfaction with the appearance of the orthodontic appliance | At the end of treatment which is expected to occur within 4 to 6 months
  Patients in both groups will be asked one question about satisfaction with the appearance of the orthodontic appliance. This question records satisfaction using a 100 mm visual analog scale (VAS). The left end of the line refers to no satisfaction (VAS=0), whereas the right end refers to maximum satisfaction (VAS=100).
Patient satisfaction with the results of the treatment | At the end of treatment which is expected to occur within 4 to 6 months
  Patients in both groups will be asked one question about their satisfaction with the treatment's results. This question records satisfaction using a 100 mm visual analog scale (VAS). The left end of the line refers to no satisfaction (VAS=0), whereas the right end refers to maximum satisfaction (VAS=100).

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Mohamad Alhafi, DDS MSc, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Nada Rajeh, DDS MSc PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University; Mohammad Younis Hajeer, DDS MSc PhD, Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, McGrath C, Hagg U. The impact of malocclusion and its treatment on quality of life: a literature review. Int J Paediatr Dent. 2006 Nov;16(6):381-7. doi: 10.1111/j.1365-263X.2006.00768.x. PMID 17014535
- [Background] Masood Y, Masood M, Zainul NN, Araby NB, Hussain SF, Newton T. Impact of malocclusion on oral health related quality of life in young people. Health Qual Life Outcomes. 2013 Feb 26;11:25. doi: 10.1186/1477-7525-11-25. PMID 23443041
- [Background] Zhang B, Huang X, Huo S, Zhang C, Zhao S, Cen X, Zhao Z. Effect of clear aligners on oral health-related quality of life: A systematic review. Orthod Craniofac Res. 2020 Nov;23(4):363-370. doi: 10.1111/ocr.12382. Epub 2020 May 13. PMID 32340082
- [Background] Azaripour A, Weusmann J, Mahmoodi B, Peppas D, Gerhold-Ay A, Van Noorden CJ, Willershausen B. Braces versus Invisalign(R): gingival parameters and patients' satisfaction during treatment: a cross-sectional study. BMC Oral Health. 2015 Jun 24;15:69. doi: 10.1186/s12903-015-0060-4. PMID 26104387
- [Background] Kara-Boulad JM, Burhan AS, Hajeer MY, Khattab TZ, Nawaya FR. Evaluation of the Oral Health-Related Quality of Life (OHRQoL) in Patients Undergoing Lingual Versus Labial Fixed Orthodontic Appliances: A Randomized Controlled Clinical Trial. Cureus. 2022 Mar 22;14(3):e23379. doi: 10.7759/cureus.23379. eCollection 2022 Mar. PMID 35371870
- [Background] Feu D, Oliveira BH, Celeste RK, Miguel JA. Influence of orthodontic treatment on adolescents' self-perceptions of esthetics. Am J Orthod Dentofacial Orthop. 2012 Jun;141(6):743-50. doi: 10.1016/j.ajodo.2011.12.025. PMID 22640676
- [Background] Palomares NB, Celeste RK, Oliveira BH, Miguel JA. How does orthodontic treatment affect young adults' oral health-related quality of life? Am J Orthod Dentofacial Orthop. 2012 Jun;141(6):751-8. doi: 10.1016/j.ajodo.2012.01.015. PMID 22640677